CLINICAL TRIAL: NCT07108049
Title: A Randomized Controlled Trial of a Couple-Based Economic Empowerment Intervention to Improve Relationship Quality and Mental Health in Three States of India
Brief Title: Strengthening Relationships and Mental Health Through a Couples-Based Economic Empowerment Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Anushree Dirangane, PhD Researcher, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TUM-EcoVi-01; ECOVI, 101115963 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2025-07-25; First posted 2025-08-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Mental Health; Empathy; Relation, Interpersonal
Keywords: Couples Intervention; Economic Empowerment; Gender Transformation; Relationship Strength; Empathy; Mental Health; GHQ-6; Cluster RCT; India; Family Economic Wellbeing; Marital Relationship Strength; Couple-based Empathy
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Let's Grow Together Intervention (Experimental): Married couples in clusters assigned to the intervention receive a structured program of six community-based sessions. Each session lasts between 2.5 and 3 hours and includes participatory activities, discussions, and exercises. All six sessions would be conducted by the same two facilitators - one male and one female. The content integrates financial literacy (e.g., household budgeting, saving practices, joint financial planning) with gender-transformative training (e.g., equitable household roles, communication skills, conflict resolution, and fostering empathy between spouses). Sessions are delivered by trained facilitators in a group setting with fifteen couples, approximately every 2-4 weeks. Some sensitive content to address economic violence context would be done in a gender segregated manner separately to encourage reflections, ensure safety and reduce defensiveness. Between sessions, SMS reminders and tips are sent to participants' mobile phones to reinforce key messages and
  Interventions: Behavioral: Let us Grow Together: Economic Wellbeing for Families
- No Structured Support (No Intervention): Married couples in clusters assigned to the control arm do not receive the special couples training during the study period. Participants in control group continue with standard activities and resources available in the community but without the structured sessions provided to the intervention arm. This control condition represents the status quo against which the added effect of the intervention can be measured. After the conclusion of the study, control clusters may be offered the intervention materials or sessions via the NGO partners in case investigators find overall positive treatment effects, ensuring ethical considerations are met.

INTERVENTIONS:
Behavioral: Let us Grow Together: Economic Wellbeing for Families — Married couples in clusters assigned to the intervention receive a structured program of six community-based sessions. Each session lasts between 2.5 and 3 hours and includes participatory activities, discussions, and exercises. All six sessions would be conducted by the same two facilitators - one male and one female. The content integrates financial literacy (e.g., household budgeting, saving practices, joint financial planning) with gender-transformative training (e.g., equitable household roles, communication skills, conflict resolution, and fostering empathy between spouses). Sessions are delivered by trained facilitators in a group setting with fifteen couples, approximately every 2-4 weeks. Some sensitive content to address economic violence context would be done in a gender segregated manner separately to encourage reflections, ensure safety and reduce defensiveness. Between sessions, SMS reminders and tips are sent to participants' mobile phones to reinforce key messages and e
  Arms: Let's Grow Together Intervention

SUMMARY:
This sub-study is part of a larger randomized controlled trial (RCT) titled Disentangling and Preventing Economic Violence against Women (ECOVI). It is conducted in rural and urban communities across Maharashtra, Andhra Pradesh, and Rajasthan, India. The sub-study evaluates the impact of a couples-based financial literacy and gender-transformative intervention on relationship strength, empathy, and mental health among married couples. Using a two-arm cluster RCT design, 150 clusters (villages or community units) are randomized to intervention or control, with ~15 husband-wife pairs per cluster (approximately 2,250 couples in total). Outcomes are measured at baseline (pre-intervention) and endline (post-intervention) approximately six months after delivery of the intervention to assess changes in perceived relationship strength, empathy (using an adapted relationship strengths and empathy scale), and mental health (General Health Questionnaire-6, GHQ-6). The study will also explore whether improvements in relationship strength and empathy mediate the intervention's effect on mental health outcomes.

DETAILED DESCRIPTION:
Studies report that couples-based programs combining financial or economic empowerment content with gender-equity and relationship-building components often yield improved relationship quality. For example, a study for low-income African-American couples describe a 20-hour workshop that significantly reduced stress and improved conflict management and relationship satisfaction at 6 months. Another study observed improved overall relationship quality among low-income couples with children, while studies from Nigeria and India document enhanced communication, trust, and joint decision-making-with adjusted relative odds for improved communication.

Interventions that combine microfinance or business training with participatory gender or relationship education report reductions in intimate partner violence-one study noted a reduction in risk by more than 50%-and improved empowerment through enhanced decision-making.

Measures of mental health and well-being, such as stress reduction and improved financial autonomy, also improved in several evaluations, although mental health outcomes appear less consistently reported than relationship outcomes. Notably, partner empathy was not an explicitly measured outcome in any study. Programs varied in intensity-from 4-8 sessions and multi-day trainings to interventions extending over 24 months-and were implemented in diverse contexts spanning low-income and rural communities in the United States, Africa, and South Asia.

This sub-study provides a focused evaluation of psychosocial outcomes within the broader "Let us Grow Together: Economic Wellbeing for Families" intervention. The main trial is designed to improve families' economic well-being through financial literacy training, while also integrating gender-transformative content to address intra-household dynamics. The sub-study specifically evaluates program impacts on marital relationship quality and mental health. It is premised on the idea that empowering couples with financial skills and promoting equitable, empathetic relationships can strengthen partner bonds and reduce psychological distress.

Participants in the intervention arm attend six structured community-based sessions for couples. These sessions blend financial literacy education (e.g. budgeting, savings, financial planning) with content on gender equity, communication, and shared decision-making. The curriculum is gender-transformative, meaning it challenges traditional gender roles and encourages empathy and cooperation between spouses. Sessions are interactive and participatory, fostering dialogue on relationship expectations, emotional support, and joint problem-solving. Between sessions, couples receive SMS text message reinforcements to encourage practice of the skills learned and to sustain engagement.

The study uses a cluster randomized controlled trial design to avoid contamination between participants. Clusters (such as villages or community centers) are randomly assigned to either the intervention or control arm by an external trial statistician. All eligible couples within intervention clusters receive the couples' sessions program, whereas couples in control clusters do not receive any structured intervention during the study period (control participants continue with services as usual). Both arms undergo identical baseline and endline assessments. The endline survey, conducted after completion of the six sessions, collects data on relationship strength, empathy, and mental health to measure changes from baseline. By comparing these changes between the intervention and control arms, the study will estimate the intervention's causal effect on the targeted outcomes.

In addition to direct outcome evaluation, an exploratory mediation analysis is planned. This analysis will test whether any improvement in mental health (GHQ-6 scores) due to the intervention occurs indirectly through enhanced relationship strength and empathy. In other words, the study will examine if the intervention's effect on participants' mental well-being is mediated by stronger couple relationships and greater spousal empathy. This will help elucidate the mechanism of impact: whether the economic and gender content improves mental health by improving how partners relate to and support each other. Findings from this sub-study will contribute to understanding the added value of integrating relationship-building and gender equity components into economic empowerment programs for families.

ELIGIBILITY:
Inclusion Criteria:

* Women: 18 - 49 years, Men: 18+
* Couples: Married and co-habitating, husband-wife pairs, who regard the selected cluster in the states Maharashtra, Andhra Pradesh, or Rajasthan of India as their primary residence for the study period.
* Consent: Both partners provide written informed consent and agree to six sessions, baseline and endline surveys, and SMS follow-ups.
* Education: Primary schooling (4th grade) complete
* Comprehension: Both partners understand the local language used in sessions.
* Availability: No plans for relocation or prolonged absence before endline.

Exclusion Criteria:

* Either partner < 18 years
* Refusal of consent or unwillingness to participate in sessions or data collection by either partner.
* Serious physical or mental condition that prevents safe, active participation (e.g., severe mental illness, debilitating disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female: 18 - 49 years, Male: 18+
Enrollment: 4500 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mental Health Scale (General Health Questionnaire - 6) | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Change in General Health Questionnaire-6 scores (psychological distress). It is scored on a scale of 0-4, where higher score indicates higher psychological distress.
  Hypothesis: Greater distress reduction (or well-being increase) in the intervention group.
Perceived Relationship Strength (PRS) | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Change in the composite Relationship Satisfaction Index (adapted for study); looking at trust, communication, mutual support, conflict resolution. The scale is scored on 1-5 scale, with higher score indicating higher perceived relationship score.
  Hypothesis: Greater improvement in the intervention group than in controls.
Relational Empathy Scale (RE) | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Adapted standardized Interpersonal Reactivity Index for Couples (emotional support, perspective-taking). The scale is scored on 1-5 scale, with higher score indicating higher empathy in relationship score.
  Hypothesis: Larger empathy gains in the intervention group.

OTHER OUTCOMES:
Proportion of the mental-health effect that is mediated | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Investigators will examine whether the intervention's impact on mental health (GHQ-6 at endline) operates partly through improvements in partner empathy and relationship strength measured at endline. Baseline levels of each construct will be adjusted for to improve precision. Empathy and relationship strength will be treated as parallel, potentially correlated mediators; investigators do not assume a temporal order between them because both are only re-measured at endline.
  Causal mediation effects will be estimated. Investigators will report (i) the indirect effect operating through endline empathy, (ii) the indirect effect operating through endline relationship strength, (iii) the remaining direct effect, and (iv) the percentage of the total treatment effect mediated by each pathway. Cluster-robust inference will be used to reflect community-level randomisation.
Moderator: Gender Norm Attitudes | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Binary classification based on baseline responses reflecting traditional vs progressive views on gender roles
Moderator: Household Economic Strain | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Self-reported household financial pressure, split at the sample median into high vs low strain.
Moderator: Residence Type | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Participant households categorized as rural or urban, based on official cluster classification.
Moderator: Living Arrangement | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Dichotomous indicator of whether the couple lives with in-laws (co-residing) or not.
Moderator: Marriage Type | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Reported as either a love marriage or an arranged marriage based on participant disclosure at baseline.
Moderator: Number of Children | T1 = baseline (prior to session 1); T2 = endline (~6 months after intervention, approx. 1.5 years after baseline))
  Categorical variable capturing whether couples have no children, 1-2 children, or 3 or more children living in the household.
  To probe possible non-linear moderation by family size, investigators will run three binary subgroup models-(i) no children, (ii) 1-2 children, (iii) ≥ 3 children-each with its own Treatment × Subgroup interaction. If sample size permits, an additional exploratory model in the Statistical Analysis Plan will treat number of children as a three-category factor (0, 1-2, 3+) or count term; results will be clearly labelled as exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Janina Steinert, Prof. Dr., Principal Investigator — Technical University of Munich
Locations (2):
- India (2):
  - 50 clusters across Maharashtra, Andhra Pradesh and Rajasthan, Mumbai, Maharashtra
  - Vayam Organisation, Noida

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. However, fully anonymized datasets may be shared with project partners and qualified researchers working on related topics (e.g., mental health and economic violence) for secondary analyses, including cross-country or pooled analyses, subject to data sharing agreements and ethical approvals.
  Timeframe: Anonymized data may be shared beginning in 2026, following primary publications.
  Access Criteria:
  Available on request upon approval by overall study PI Prof. Dr. Steinert

REFERENCES:
- [Background] Falconier, M. K., Kim, J., & Lachowicz, M. J. (2023). Together-A couples' program integrating relationship and financial education: A randomized controlled trial. Journal of Social and Personal Relationships, 40(1), 333-359. https://doi.org/10.1177/02654075221118816
- [Background] Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007 Dec;21(4):572-83. doi: 10.1037/0893-3200.21.4.572. PMID 18179329
- [Background] Imai K, Keele L, Tingley D. A general approach to causal mediation analysis. Psychol Methods. 2010 Dec;15(4):309-34. doi: 10.1037/a0020761. PMID 20954780
- [Background] Ismayilova L, Karimli L, Gaveras E, To-Camier A, Sanson J, Chaffin J, Nanema R. An Integrated Approach to Increasing Women's Empowerment and Reducing Domestic Violence: Results of a Cluster-Randomized Controlled Trial in a West African Country. Psychol Violence. 2018 Jul;8(4):448-459. doi: 10.1037/vio0000136. Epub 2017 Aug 7. PMID 34790432
- [Background] John NA, Adebayo A, Boychuk NA, OlaOlorun F. Intimate partner violence (IPV) prevention using a cross-sectoral couple-based intervention: results from a cluster randomised control trial in Ibadan, Nigeria. BMJ Glob Health. 2022 Feb;7(2):e007192. doi: 10.1136/bmjgh-2021-007192. PMID 35140139
- [Background] Kim JC, Watts CH, Hargreaves JR, Ndhlovu LX, Phetla G, Morison LA, Busza J, Porter JD, Pronyk P. Understanding the impact of a microfinance-based intervention on women's empowerment and the reduction of intimate partner violence in South Africa. Am J Public Health. 2007 Oct;97(10):1794-802. doi: 10.2105/AJPH.2006.095521. Epub 2007 Aug 29. PMID 17761566
- [Background] Moore, Q., Wood, R. G., & Wu, A. Y. (2023). Impacts of healthy marriage and relationship education with integrated economic stability services. Family Relations, 72(4), 1422-1440. https://doi.org/10.1111/fare.12877
- [Background] Peloquin K, Lafontaine MF. Measuring empathy in couples: validity and reliability of the Interpersonal Reactivity Index for couples. J Pers Assess. 2010 Mar;92(2):146-57. doi: 10.1080/00223890903510399. PMID 20155564
- [Background] Raj A, Ghule M, Johns NE, Battala M, Begum S, Dixit A, Vaida F, Saggurti N, Silverman JG, Averbach S. Evaluation of a gender synchronized family planning intervention for married couples in rural India: The CHARM2 cluster randomized control trial. EClinicalMedicine. 2022 Mar 5;45:101334. doi: 10.1016/j.eclinm.2022.101334. eCollection 2022 Mar. PMID 35274093
- [Background] Rao KN, Begum S, Siddappa K, Ravindra K. Validity of a 6-item version of general health questionnaire (g.h.q.) in the hands of a non - psychiatrist. Indian J Psychiatry. 1992 Apr;34(2):145-7. PMID 21776115
- See also: Project Website — https://sites.google.com/view/ecovi-project/home

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT07108049/Prot_SAP_000.pdf